CLINICAL TRIAL: NCT01852136
Title: Clinical Evaluation of the BD NEXT (Extra Thin Wall Pen Needles) Compared to the Currently Marketed Pen Needles
Brief Title: Clinical Evaluation of BD NEXT Pen Needle
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: DBC-11-NEXXT01
Record Dates: First submitted 2013-05-09; First posted 2013-05-13 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
Keywords: pen needle; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- NEXT 31G x 5mm: Subjects will use their current pen needle or the BD NEXT 31G x 5mm pen needle for approximately one week (Period 1). The alternate pen needle will be used for one week in Period 2.
  Interventions: Device: BD NEXT 31G x 5 mm pen needle
- NEXT 31G x 8mm: Subjects will use their current pen needle or the BD NEXT 31G x 8mm pen needle for approximately one week (Period 1). The alternate pen needle will be used for one week in Period 2.
  Interventions: Device: BD NEXT 31G x 8mm pen needle
- NEXT 32G x 4mm: Subjects will use their current pen needle or the BD NEXT 32G x 4mm pen needle for approximately one week (Period 1). The alternate pen needle will be used for one week in Period 2.
  Interventions: Device: BD NEXT 32G x 4mm pen needle

INTERVENTIONS:
Device: BD NEXT 31G x 5 mm pen needle — Each pen needle type will be used for approximately one week. Subjects will use their current pen injector device.
  Groups: NEXT 31G x 5mm
Device: BD NEXT 31G x 8mm pen needle — Each pen needle type will be used for approximately one week. Subjects will use their current pen injector device.
  Groups: NEXT 31G x 8mm
Device: BD NEXT 32G x 4mm pen needle — Each pen needle type will be used for approximately one week. Subjects will use their current pen injector device.
  Groups: NEXT 32G x 4mm

SUMMARY:
This prospective, multi-center, 2 period cross-over study is designed to determine if people who use injection pens for subcutaneous medication delivery prefer the BD NEXT pen needle (PN) in comparison with currently marketed pen needles of the same or similar gauge and length. Subjects will use the investigational (BD NEXT) PN and their usual conventional PN each for one week in a randomly assigned sequence, and will be asked to evaluate and compare characteristics of the BD NEXT pen needle versus their usual pen needle when used for all their pen injections performed at home. Since injection experience may vary according to the type of pen device used, equal numbers of subjects will be recruited who are users of three of the most commonly used insulin pen injectors.

DETAILED DESCRIPTION:
Using their usual insulin doses, pen and injection routine, subjects will be asked to compare two different pen needles (PNs) of corresponding gauge (GA) and length, one being the investigational (extra thin wall) pen needle and the other being their most often, currently used pen needle. Based on their current pen needle gauge and length, subjects will be assigned to the BD NEXT pen needle with the most comparable gauge (G) and length, in millimeters (mm). The three possible sizes are BD NEXT 32G x 4mm pen needle, BD NEXT 31G x 5mm pen needle, or BD NEXT 31G x 8 mm pen needle.

Both study pen needles will be used by the subject on the same pen device/insulin brand. If subjects are using two different pens, comparison data will be collected for both pen devices.

Each subject will participate in three study visits over the course of approximately 3 weeks. Study conduct will include two in-home use study periods each lasting approximately (1) one week.

During Visit 1, after subjects are enrolled and assigned to a pen device group, subjects will be randomly assigned to use the BD NEXT or their usual PN for use during a 1 week home use period (Period 1). After approximately 1 week, at Visit 2, subjects will be crossed-over to the other study PN per the randomization schedule.

After approximately 1 week of home use with the second study PN (Period 2), at Visit 3, subjects will be asked to complete Visual Analog Scales (VAS) and answer questions comparing their injection experiences with the two different PNs.

The primary and secondary objectives will be assessed for all pen users combined. In addition, preference, thumb force, and confidence in full dose delivery will be compared among the subsets of subjects using each of the following pen devices: sanofi-aventis SoloSTAR®, Lilly KwikPen™, Novo Nordisk FlexPen®. In order to achieve a minimum of 60 evaluable subjects in each of these pen user groups approximately 210 subjects will be enrolled (70 subjects per pen group).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 1 or Type 2 diabetes.
* Currently self-injects insulin with a pen device at least once daily, and doing so for at least two months prior to enrollment.
* One or more daily insulin doses injected with the pen device must be > 10 units
* The insulin pen being used by the subject for the daily dose of > 10 units must be one of the three currently marketed pens: sanofi-aventis SoloSTAR, Lilly KwikPen, or Novo Nordisk FlexPen
* Using a pen needle that is either 4, 5, 6, or 8 mm length, and either 31 or 32 gauge.
* Willing to use the assigned study needles for all pen injections (including insulin and any other pen-based medications).
* Willing to keep their diabetes medications, diet, and exercise the same during the study.
* Able to read, write and follow instructions in English.
* Able and willing to provide informed consent.
* The subject may also be using syringe and vial for some insulin doses, provided that at least one injection per day is done with an insulin pen and pen needle and is > 10 units.

Exclusion Criteria:

* Have previous knowledge of the details of this study or investigational products.
* Current status or history of a medical condition that would contraindicate treatment with study products or other conditions which, in the opinion of the Principal Investigator or Sub-Investigator, would place the subject at risk or have the potential to confound interpretation of the study results (e.g., recent history of ketoacidosis, hypoglycemic unawareness, etc.).
* Currently participating in any other clinical investigation that conflicts with this one, or who have participated in a study with the same indication within the prior 30 days that the Principal Investigator or Sub-Investigator believes will conflict with outcomes or ability of the subject to complete all activities required in this study.
* Currently using either the Pic Indolor (Artsana) Insupen Sensitive 8 mm X 32G pen needle or the Pic Indolor (Artsana) Insupen Sensitive 6mm X 32G pen needle.
* History of intravenous drug use (self-reported).
* Employee, contractor or consultant to any company that manufactures pen needles, including BD.
* Pregnant (self-reported).

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Overall Pen Needle Preference | End of Period 2, after using each assigned pen needle for 1 week
  The primary objective was assessed using a 15 cm VAS. A vertical line drawn to the left of the VAS center mark indicates that the Study Period 1 PN was preferred more than the Study Period 2 PN. Those PNs will be scored in (-) mm (maximum score -75 mm). A vertical line drawn to the right of the VAS center mark indicates that the Study Period 2 PN was preferred more than the Study Period 1 PN. Those PNs will be scored in (+) mm (maximum score +75 mm). The sign of the reading will be adjusted depending on which PN was tested first, so that the readings will represent relative differences of Investigational PN and Current PN, with positive scores indicating preference for the investigational PN. The difference between the BD NEXT PN and subject's usual PN is statistically significant if the entire 95% confidence interval (CI) is either positive (BD NEXT preferred) or negative (current PN preferred) with respect to preference assessment.

SECONDARY OUTCOMES:
Relative perceived thumb force | End of Period 2, after using each assigned PN for 1 week
  Using a similar 15 cm VAS as for the primary objective, subjects will be asked to compare the BD NEXT with their usual marketed pen needle to assess relative perceived thumb force to deliver insulin. The VAS will be measured as described for the primary objective.
Confidence in full dose delivery of insulin | End of Period 2, after using each assigned PN for 1 week
  Using a 15 cm VAS, at the final study visit subjects will be asked to compare the BD NEXT with their usual marketed pen needle to assess relative confidence in a full dose delivery of insulin. The VAS will be measured as described for the primary objective.
Perceived injection time to deliver full dose of insulin | End of Period 2, after using each assigned PN for 1 week
  Subjects will use a 15 cm VAS to compare the BD NEXT with their usual marketed pen needle to assess relative perceived injection time to deliver the full dose. The VAS will be measured as described for the primary objective.
Pen user group subset comparisons | End of Period 2, after using each assigned PN for 1 week
  The VAS responses for preference, thumb force required to deliver insulin and confidence in delivering a full dose by subjects when using the BD NEXT pen needle in comparison with their usual pen needles were compared among the subsets of subjects using each of the following pen devices: sanofi-aventis SoloSTAR®, Lilly KwikPen™, and Novo Nordisk FlexPen®.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence J Hirsch, MD, Study Director — BD Medical-Diabetes Care
Locations (5):
- United States (4):
  - Physicians Research Center, Toms River, New Jersey
  - Mountain Diabetes and Endocrine Center, Asheville, North Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Corporation Lane Internal Medicine and Research Center, Virginia Beach, Virginia
- LMC Endocrinology Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aronson R, Gibney MA, Oza K, Berube J, Kassler-Taub K, Hirsch L. Insulin pen needles: effects of extra-thin wall needle technology on preference, confidence, and other patient ratings. Clin Ther. 2013 Jul;35(7):923-933.e4. doi: 10.1016/j.clinthera.2013.05.020. Epub 2013 Jun 20. PMID 23790553